CLINICAL TRIAL: NCT05745766
Title: Evaluation of the Diagnostic Accuracy of Cone-beam Computed Tomography (CBCT) Imaging Compared to the Two-dimensional (2D) Methods in the 3D Localization and Assessment of Maxillary Impacted Canines: A Surgical-exposure-based Study
Brief Title: 2D Versus 3D Radiographs in the Localization of Upper Impacted Canines
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Ortho-01-2023
Record Dates: First submitted 2023-02-13; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Impacted Canines
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Canines assessed using 2D images: The 2D-based assessments of the impacted maxillary canine.
  Interventions: Other: Panoramic and lateral cephalometric radiography
- Canines assessed using 3D images: The 3D-based assessments of the impacted maxillary canine.
  Interventions: Other: Cone beam computed tomography
- Canines assessed intra-operatively or post-operatively: The gold standard-based assessments are based on surgical exposure.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Panoramic and lateral cephalometric radiography — The 2D-based assessments of the impacted maxillary canine will be achieved using panoramic and lateral cephalometric radiographs.
  Groups: Canines assessed using 2D images
Other: Cone beam computed tomography — The 3D-based assessments of the impacted maxillary canine will be achieved using a cone beam computed tomography (CBCT) image.
  Groups: Canines assessed using 3D images
Other: Surgery — The surgical exposure will be accomplished, and the impacted maxillary canine will be assessed by a direct vision.
  Groups: Canines assessed intra-operatively or post-operatively

SUMMARY:
Seventeen patients diagnosed with the extraction-based treatment of impacted maxillary canines will be included in this study. Each patient will undergo conventional 2D radiography including panoramic, and lateral cephalometric, in addition to 3D imaging by cone beam computed tomography (CBCT) images.

A set of variables will be evaluated on 2D and 3D images by a panel of assessors and then these results will be compared with the gold standard which will be established based on surgical detection and direct visualization of the impacted canine.

DETAILED DESCRIPTION:
After taking the radiographic records, the impacted maxillary canines will be surgically exposed under local anesthesia where a full-thickness flap will be elevated from the buccal or palatal according to the initial radiographic diagnosis.

After cleaning the work yard to achieve good visibility, the pre-extraction parameters will be recorded which will be included labiopalatal position, mesiodistal position, and vertical position of the canine cusp, in addition to ankyloses of the impacted maxillary canine, proximity to the adjacent teeth, resorption of the adjacent incisors induced by the impacted maxillary canine, and bony coverage of the canine crown.

This will be followed by the extraction of the upper impacted canine and the recording of the post-extraction parameters, which will include the shape and the root apex development of the extracted canine. The pre- and post-extraction readings will be deemed the gold standard which will be compared to the 2D- and 3D-based assessments of the assessors.

Assessment sessions will be divided into two sessions with a one-week break in between. The first session will be devoted to the evaluation of the 2D image sets, while the second one will be to the evaluation of the 3D images.

Before beginning the assessment, the assessors will be subjected to a set of instructions and clarifications, including a set of graphs that help each assessor to accurately identify each variable, in addition to an oral explanation of some points so that the assessor will not fall into doubt when evaluating the radiographs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from both gender (Male and female), Age range: 14-27 years.
2. Unilateral impaction of the maxillary canines requiring surgical extraction.
3. Non-syndromic patients without any pathology of the maxillofacial region (benign or malignant tumor, cleft lip or cleft palate, trauma)
4. Patients with a set of panoramic and lateral cephalometric images, in addition to CBCT radiograph (CBCT is indicated for treatment planning)
5. The time period between taking the radiological records and undergoing the surgical intervention does not exceed four weeks

Exclusion Criteria:

1. Patients who had a systemic disorder, cleft lip/cleft palate, craniofacial syndrome, traumatic injury, and congenital number anomaly.
2. Patients had previous orthodontic treatment.

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with impacted canines. These canines should be located unilaterally. The orthodontic decision should include the removal of these impacted canines in the course of orthodontic treatment.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Labiopalatal position of the canine cusp | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed relative to the adjacent teeth based on classification into three categories: 1-Labial, 2-In situ, 3- Palatal
Mesiodistal position of the canine cusp | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on classification into five sectors: Section (B') From the distal margin of the central incisor to the midline of the Palatine. Section (B) Between the mesial and distal margins of the lateral incisor on the same side of the impaction. Section (A) Between the distal of the lateral incisor and the mesial of the 1st premolar on the same side of the impaction. Section (C) Between the mesial and distal margins of the 1st premolar on the same side of the impaction. Section (C') Between the distal of the 1st premolar and the distal of the 2nd premolar.
The vertical position of the canine cusp | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on classification into three categories: 1-The cervical third, 2-The middle third, 3-The apical third
Ankylosis of the impacted maxillary canine | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on periodontal ligament distance (the canine root will be considered ankylosis if the periodontal ligament distance is equal to zero)
Proximity to the adjacent teeth | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on contact with the root of the adjacent incisor (the canine will be considered in contact when the space by 0 mm or less than 0.5 mm)
Resorption of the adjacent incisors induced by the impacted canine | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on the presence or absence of resorption in the adjacent teeth.
Bony coverage of the impacted maxillary canine | The assessment will be performed after the surgical exposure of the impacted maxillary canine and "during surgery", i.e., after 10 minutes of the surgical exposure.
  Assessment will be performed based on the classification of the bony coverage amount of the impacted canine crown into: 1- Completely covered with bone, 2- Partially covered with bone, 3- Uncovered
The shape of the extracted canine | The assessment will be performed after the extraction of the impacted maxillary canine, i.e., immediately following surgery
  Assessment will be performed based on the angle between the long axis of both the root and the crown and it will be classified into: 1-Straight (0°-10°), 2-Mildly curved (10°-30°), 3-Severe curved (>30°)
Root apex closure of the extracted canine | The assessment will be performed after the extraction of the impacted maxillary canine, i.e., immediately following surgery
  Assessment will be performed based on classification into two categories: 1-Open apex, 2- Closed apex
Diagnostic accuracy, sensitivity, and specificity | The assessment will be performed after the extraction of the impacted maxillary canine, i.e., immediately following surgery
  Values of the parameters were assessed using CBCT and 2D radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Shaweesh, DDS MSc, Principal Investigator — Department of Oral and Maxillofacial Surgery, Damascus University, Syria; Doa'a Tahseen Alfailany, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y. Hajeer, DDS MSc PhD, Study Director — Department of orthodontics, Damascus University, Syria; Bassel Brad, DDS MSc PhD, Study Chair — Department of Oral and Maxillofacial Surgery, Damascus University, Syria
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Damascus Faculty of Dentistry, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker L, Enciso R, Mah J. Three-dimensional localization of maxillary canines with cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2005 Oct;128(4):418-23. doi: 10.1016/j.ajodo.2004.04.033. PMID 16214621
- [Background] Alqerban A, Storms AS, Voet M, Fieuws S, Willems G. Early prediction of maxillary canine impaction. Dentomaxillofac Radiol. 2016;45(3):20150232. doi: 10.1259/dmfr.20150232. Epub 2015 Dec 18. PMID 26683426
- [Background] Al-Homsi HK, Hajeer MY. An Evaluation of Inter- and Intraobserver Reliability of Cone-beam Computed Tomography- and Two Dimensional-based Interpretations of Maxillary Canine Impactions using a Panel of Orthodontically Trained Observers. J Contemp Dent Pract. 2015 Aug 1;16(8):648-56. doi: 10.5005/jp-journals-10024-1736. PMID 26423501
- [Background] Botticelli S, Verna C, Cattaneo PM, Heidmann J, Melsen B. Two- versus three-dimensional imaging in subjects with unerupted maxillary canines. Eur J Orthod. 2011 Aug;33(4):344-9. doi: 10.1093/ejo/cjq102. Epub 2010 Dec 3. PMID 21131389
- [Background] Hajeer MY, Al-Homsi HK, Alfailany DT, Murad RMT. Evaluation of the diagnostic accuracy of CBCT-based interpretations of maxillary impacted canines compared to those of conventional radiography: An in vitro study. Int Orthod. 2022 Jun;20(2):100639. doi: 10.1016/j.ortho.2022.100639. Epub 2022 May 21. PMID 35606269